CLINICAL TRIAL: NCT04024501
Title: A Randomised, Single-dose, 5-period, 5-treatment, Crossover Study to Assess the Relative Bioavailability of 3 Different Extended-release Formulations of Verinurad in Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability of 3 Different Formulations Under Fasted and Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5495C00005
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Chronic Kidney Disease
Keywords: URAT1 inhibitor; Uric acid transporter 1; Verinurad; Crossover study; Relative bioavailability; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment 1 (Experimental): During this treatment period, healthy participants will receive 1 x 12 mg verinurad ER8 capsule formulation in fasted state.
  Interventions: Drug: Verinurad ER8 capsule formulation (fasted)
- Treatment 2 (Experimental): During this treatment period, healthy participants will receive 2 x 6 mg verinurad A-capsule formulation in fasted state.
  Interventions: Drug: Verinurad A-capsule formulation (fasted)
- Treatment 3 (Experimental): During this treatment period, healthy participants will receive 2 x 6 mg verinurad A-capsule formulation in fed state.
  Interventions: Drug: Verinurad A-capsule formulation (fed)
- Treatment 4 (Experimental): During this treatment period, healthy participants will receive 2 x 6 mg verinurad B-capsule formulation in fasted state.
  Interventions: Drug: Verinurad B-capsule formulation (fasted)
- Treatment 5 (Experimental): During this treatment period, healthy participants will receive 2 x 6 mg verinurad B-capsule formulation in fed state.
  Interventions: Drug: Verinurad B-capsule formulation (fed)

INTERVENTIONS:
Drug: Verinurad ER8 capsule formulation (fasted) — Each participant will receive single-dose treatment of 12 mg verinurad ER8 capsule with 240 mL water, following an overnight fast of at least 10 hours.
  Arms: Treatment 1
Drug: Verinurad A-capsule formulation (fasted) — Each participant will receive single-dose treatment of 12 mg verinurad A-capsule with 240 mL water, following an overnight fast of at least 10 hours.
  Arms: Treatment 2
Drug: Verinurad A-capsule formulation (fed) — Each participant will receive single dose treatment of 12 mg verinurad A-capsule with 240 mL water, following a high-fat, high-calorie breakfast (after the overnight fast).
  Arms: Treatment 3
Drug: Verinurad B-capsule formulation (fasted) — Each participant will receive single-dose treatment of 12 mg verinurad B-capsule with 240 mL water, following an overnight fast of at least 10 hours.
  Arms: Treatment 4
Drug: Verinurad B-capsule formulation (fed) — Each participant will receive single dose treatment of 12 mg verinurad B-capsule with 240 mL water, following a high-fat, high-calorie breakfast (after the overnight fast).
  Arms: Treatment 5

SUMMARY:
This study is intended to assess the relative bioavailability between the (extended-release) ER8 capsule formulation (the formulation that is currently used for verinurad development) given under fasted conditions and 2 new capsule formulations of verinurad (A-capsule and B-capsule) given under fed or fasted conditions. All three capsules target an 8-hour release profile (extended-release). The highest dose (12 mg) currently tested in participants will be tested in this study. The study is designed to provide information to optimize the verinurad part of a fixed dose combination capsule to be used in future development.

DETAILED DESCRIPTION:
This study will be a randomised, open-label, single-dose, 5-period, 5-treatment, crossover study in healthy male and female participants, performed at a single study centre. This study is intended to assess the relative bioavailability between the ER8 capsule formulation (the formulation that is currently used for verinurad development) given under fasted conditions and 2 new capsule formulation of verinurad (A-capsule and B-capsule) given under fed or fasted conditions. All three capsules target an 8-hour release profile (extended-release). The highest dose (12 mg) currently tested in participants will be tested in this study. The study is designed to provide information to optimize the verinurad part of a fixed dose combination capsule to be used in future development. The study will comprise: a screening period of maximum 28 days; five treatment periods during which participants will be resident from the morning of the day before dosing with verinurad (Day -1) until at least 72 hours after dosing; discharged on the morning of Day 4 of each Treatment Period; and a follow-up Visit within 7 to 14 days after the last administration of verinurad. There will be a minimum washout period of 5 days between each dose administration. A total of 25 healthy male and female participants will be randomised into this study. Each participant will receive five single-dose treatments of 12 mg verinurad with 240 mL water, following an overnight fast of at least 10 hours. Participants will follow an overnight fast of at least 10 hours before the dosing procedures: for the fed dosing, a high-fat, high-calorie standard breakfast will be served 30 minutes before the planned administration of verinurad to be consumed in full at least 5 minutes before dosing; for the fasted dosing, no breakfast will be served. A meal can be given 4 hours after administration of verinurad for both dosing states. The duration of the study is expected to be approximately 9 weeks for each individual participant (including the 28-day screening period).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and female participants aged 18 to 50 years with suitable veins for cannulation or repeated venepuncture.
3. Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg.
4. Females must have a negative pregnancy test at screening and on admission to the unit and must be:

(1) not pregnant or currently lactating or breastfeeding. (2) of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria: (i) postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range (FSH levels > 40 IU/mL).

(ii) documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

(3) OR if of childbearing potential must be willing to use an acceptable method of contraception to avoid pregnancy for the entire study period.

Exclusion Criteria:

1. History of gout or any clinically significant disease or disorder which, in the opinion of the Principal Investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of verinurad.
3. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
4. Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results as judged by the Investigator at screening and first admission, including: (1) Alanine aminotransferase (ALT) > 1.5 x upper limit of normal (ULN), (2) Aspartate aminotransferase (AST) > 1.5 x ULN, (3) Bilirubin (total) > 1.5 x ULN, (4) Gamma glutamyl transpeptidase (GGT) > 1.5 x ULN. (5) If any of these tests are out-of-range, the tests can be repeated once.
5. Any clinically significant abnormal findings in vital signs at the Screening Visit and/or admission to the Clinical Unit, including, but not limited to, any of the following:

(1) Heart rate (resting, supine) < 50 beats per minute (bpm) or > 85 bpm, (2) Systolic BP < 90 mmHg or > 140 mmHg and/or diastolic BP < 50 mmHg or > 90 mmHg sustained for > 10 min while resting in a supine position.

6. Any clinically significant abnormalities on 12-lead Electrocardiogram (ECG) at the Screening Visit, including, but not limited to any of the following:

1. ECG interval measured from the onset of the QRS complex to the end of the T wave (QT) interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms or < 340 ms or family history of long QT syndrome,
2. Any significant arrhythmia,
3. Conduction abnormalities:
4. Clinically significant PR (PQ) interval prolongation (> 240 ms); intermittent second or third degree atrioventricular (AV) block, or AV dissociation,
5. Complete bundle branch block and/or QRS duration > 120 ms. 7. Any positive result at the Screening Visit for serum hepatitis B surface antigen or antiHBc antibody, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

8. Suspicion or known Gilbert's and/or Lesch-Nyhan syndrome. 9. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for women.

10. Has received another new chemical entity (defined as a compound which has not been approved for marketing in the US) within 30 days or at least 5 half-lives (whichever is longer) of the first administration of verinurad in this study.

11. Participants who have previously received verinurad. 12. Plasma donation within 1 month of screening or any blood donation/loss of more than 500 mL during the 3 months prior to the Screening Visit.

13. Participants who are pregnant, lactating or planning to become pregnant. 14. History of severe allergy/hypersensitivity or ongoing clinically relevant allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to verinurad.

15. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.

16. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the PI. Excessive intake of caffeine defined as regular consumption of more than 600 mg of caffeine per day (e.g., > 5 cups of coffee) or would likely be unable to refrain from the use of caffeine containing beverages during confinement at the investigational site.

17. Positive screen for drugs of abuse or cotinine (nicotine) at the Screening Visit or positive screen for alcohol, drugs of abuse and cotinine on each admission to the study centre.

18. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of verinurad.

19. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of verinurad or longer if the medication has a long half-life. The use of hormonal contraception therapy and hormonal replacement therapy for females are permitted.

20. Any AstraZeneca, PAREXEL or study site employee or their close relatives. 21. Participants who cannot communicate reliably with the PI and/or is not able to read, speak and understand the German language.

22. Judgment by the PI that the participant should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

23. Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

24. Participants with any special dietary restrictions such as participants that are lactose intolerant or are vegetarians/vegans.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

REFERENCES:
- See also: redacted CSP and SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00005&attachmentIdentifier=47483f56-39b2-4098-ae5a-75c4996ee4eb&fileName=d5495c00005_clinical_study_protocol_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects signed and dated the informed consent form (ICF) before any study procedures were performed.
Pre-assignment Details: The study included a Screening Period of maximum 28 days.
Groups:
- Overall-All Subjects: All subjects were randomized into 5-period, 5-treatment, crossover study to receive a single oral dose of 12 mg verinurad:
  * Treatment 1: 1 x 12 mg verinurad ER8 capsule formulation, fasted.
  * Treatment 2: 2 x 6 mg verinurad A-capsule formulation, fasted.
  * Treatment 3: 2 x 6 mg verinurad A-capsule formulation, fed.
  * Treatment 4: 2 x 6 mg verinurad B-capsule formulation, fasted.
  * Treatment 5: 2 x 6 mg verinurad B-capsule formulation, fed.
Period: Overall Study
Arm/Group | Overall-All Subjects
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall-All Subjects
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time Curve From Zero to Infinity (AUC)
Description: To evaluate the relative bioavailability between the A-capsule and B-capsule formulations under both fed and fasted conditions with the ER8 capsule formulation under fasted conditions and with each other under the same food conditions.
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: The PK analysis set consisted of all subjects in the safety analysis set for whom at least 1 of the primary PK parameters could be calculated, and who had no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Treatment 1: 1 x 12 mg ER8 Capsule Fasted: During this treatment period, healthy participants will receive 1 x 12 mg verinurad ER8 capsule formulation in fasted state.
- Treatment 2: 2 x 6 mg A-capsule Fasted: During this treatment period, healthy participants will receive 2 x 6 mg verinurad A-capsule formulation in fasted state.
- Treatment 3: 2 x 6 mg A-capsule Fed: During this treatment period, healthy participants will receive 2 x 6 mg verinurad A-capsule formulation in fed state.
- Treatment 4: 2 x 6 mg B-capsule Fasted: During this treatment period, healthy participants will receive 2 x 6 mg verinurad B-capsule formulation in fasted state.
- Treatment 5: 2 x 6 mg B-capsule Fed: During this treatment period, healthy participants will receive 2 x 6 mg verinurad B-capsule formulation in fed state.
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng*h/mL | 171.3 (47.60) | 167.5 (33.72) | 87.14 (65.84) | 149.0 (39.78) | 150.2 (42.57)
Statistical Analysis 1: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 2: 2 x 6 mg A-capsule Fasted; Pairwise comparison: Treatment 2/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 22; Geometric Mean ratio = 106.20, 90% CI 2-sided [91.73 to 122.96]
Statistical Analysis 2: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 3: 2 x 6 mg A-capsule Fed; Pairwise comparison: Treatment 3/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 22; Geometric mean ratio = 50.02, 90% CI 2-sided [42.34 to 59.10]
Statistical Analysis 3: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 3: 2 x 6 mg A-capsule Fed; Pairwise comparison: Treatment 3/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 15; Geometric mean ratio = 47.10, 90% CI 2-sided [39.85 to 55.68]
Statistical Analysis 4: Comparison: Treatment 3: 2 x 6 mg A-capsule Fed vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 3/Treatment 4; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 15; Geometric mean ratio = 58.40, 90% CI 2-sided [49.49 to 68.92]
Statistical Analysis 5: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 4/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 21; Geometric mean ratio = 85.65, 90% CI 2-sided [73.78 to 99.43]
Statistical Analysis 6: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 4/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 21; Geometric mean ratio = 80.65, 90% CI 2-sided [69.48 to 93.62]
Statistical Analysis 7: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 21; Geometric mean ratio = 89.88, 90% CI 2-sided [77.61 to 104.09]
Statistical Analysis 8: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 21; Geometric mean ratio = 84.64, 90% CI 2-sided [72.94 to 98.20]
Statistical Analysis 9: Comparison: Treatment 3: 2 x 6 mg A-capsule Fed vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 3; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 21; Geometric mean ratio = 179.68, 90% CI 2-sided [151.57 to 212.99]
Statistical Analysis 10: Comparison: Treatment 4: 2 x 6 mg B-capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 4; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 21; Geometric mean ratio = 104.94, 90% CI 2-sided [90.18 to 122.11]

2. Primary Outcome: AUC From Time 0 to the Last Quantifiable Concentration (AUC0-t) for the Analysis of PK Parameter
Description: as for outcome 1
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng*h/mL | 166.8 (47.57) | 167.5 (35.96) | 67.04 (80.37) | 128.5 (49.29) | 139.6 (44.36)
Statistical Analysis 1: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 2: 2 x 6 mg A-capsule Fasted; Pairwise comparison: Treatment 2/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 25; Geometric mean ratio = 100.39, 90% CI 2-sided [84.94 to 118.65]
Statistical Analysis 2: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 3: 2 x 6 mg A-capsule Fed; Pairwise comparison: Treatment 3/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 41.26, 90% CI 2-sided [34.74 to 49.00]
Statistical Analysis 3: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 3: 2 x 6 mg A-capsule Fed; Pairwise comparison: Treatment 3/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 41.10, 90% CI 2-sided [34.61 to 48.81]
Statistical Analysis 4: Comparison: Treatment 3: 2 x 6 mg A-capsule Fed vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 3/Treatment 4; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 53.55, 90% CI 2-sided [45.09 to 63.59]
Statistical Analysis 5: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 4/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 25; Geometric mean ratio = 77.05, 90% CI 2-sided [65.19 to 91.06]
Statistical Analysis 6: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 4/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 25; Geometric mean ratio = 76.75, 90% CI 2-sided [64.94 to 90.71]
Statistical Analysis 7: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 84.23, 90% CI 2-sided [70.93 to 100.03]
Statistical Analysis 8: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 83.90, 90% CI 2-sided [70.65 to 99.64]
Statistical Analysis 9: Comparison: Treatment 3: 2 x 6 mg A-capsule Fed vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 3; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 204.16, 90% CI 2-sided [171.22 to 243.42]
Statistical Analysis 10: Comparison: Treatment 4: 2 x 6 mg B-capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 4; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 109.32, 90% CI 2-sided [92.06 to 129.83]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for the Analysis of PK Parameter
Description: as for outcome 1
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng/mL | 25.51 (53.66) | 31.88 (62.41) | 8.243 (81.12) | 23.39 (66.08) | 17.02 (54.00)
Statistical Analysis 1: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 2: 2 x 6 mg A-capsule Fasted; Pairwise comparison: Treatment 2/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 25; Geometric mean ratio = 124.99, 90% CI 2-sided [101.09 to 154.54]
Statistical Analysis 2: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 3: 2 x 6 mg A-capsule Fed; Pairwise comparison: Treatment 3/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 33.77, 90% CI 2-sided [27.15 to 42.01]
Statistical Analysis 3: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 3: 2 x 6 mg A-capsule Fed; Pairwise comparison: Treatment 3/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 27.02, 90% CI 2-sided [21.72 to 33.61]
Statistical Analysis 4: Comparison: Treatment 3: 2 x 6 mg A-capsule Fed vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 3/Treatment 4; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 36.84, 90% CI 2-sided [29.61 to 45.82]
Statistical Analysis 5: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 4/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 25; Geometric mean ratio = 91.69, 90% CI 2-sided [74.15 to 113.36]
Statistical Analysis 6: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 4: 2 x 6 mg B-capsule Fasted; Pairwise comparison: Treatment 4/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 25; Geometric mean ratio = 73.36, 90% CI 2-sided [59.33 to 90.70]
Statistical Analysis 7: Comparison: Treatment 1: 1 x 12 mg ER8 Capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 1; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 67.62, 90% CI 2-sided [54.37 to 84.12]
Statistical Analysis 8: Comparison: Treatment 2: 2 x 6 mg A-capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 2; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 54.11, 90% CI 2-sided [43.50 to 67.30]
Statistical Analysis 9: Comparison: Treatment 3: 2 x 6 mg A-capsule Fed vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 3; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 200.23, 90% CI 2-sided [160.15 to 250.32]
Statistical Analysis 10: Comparison: Treatment 4: 2 x 6 mg B-capsule Fasted vs Treatment 5: 2 x 6 mg B-capsule Fed; Pairwise comparison: Treatment 5/Treatment 4; Test type: Other; Mixed Model Analysis; The number of subjects in this analysis: 23; Geometric mean ratio = 73.76, 90% CI 2-sided [59.30 to 91.75]

4. Secondary Outcome: AUC From Time 0 to 24 Hours Post Dose (AUC0-24) for the Analysis of PK Parameter
Description: To examine the PK profiles of verinurad when administered as the 3 different capsule formulations under fasted conditions.
Time Frame: Pre-dose and up to 24-hours Post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng*h/mL | 132.6 (48.40) | 138.5 (39.67) | 54.85 (80.02) | 102.9 (54.45) | 110.6 (47.83)

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for the Analysis of PK Parameter
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Hour | 4.98 [3.00 to 8.00] | 4.98 [2.98 to 6.02] | 5.00 [3.00 to 10.00] | 4.00 [2.00 to 6.00] | 7.98 [4.00 to 12.00]

6. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz) for the Analysis of PK Parameter
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Hour | 14.02 (4.732) | 13.61 (5.748) | 13.42 (5.549) | 14.36 (5.477) | 12.40 (5.038)

7. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (CL/F) for the Analysis of PK Parameter
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre/hour
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Litre/hour | 77.86 (42.15) | 75.43 (25.71) | 160.5 (86.96) | 86.26 (32.22) | 87.10 (41.78)

8. Secondary Outcome: Mean Residence Time of the Unchanged Drug in the Systemic Circulation From Zero to Infinity (MRT) for the Analysis of PK Parameter
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Hour | 16.98 (4.006) | 15.52 (5.843) | 17.43 (4.974) | 16.61 (6.049) | 18.28 (4.841)

9. Secondary Outcome: Time of Last Quantifiable Plasma Concentration (Tlast) for the Analysis of PK Parameter
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Hour | 71.65 [47.67 to 72.93] | 48.47 [36.00 to 72.05] | 47.97 [35.97 to 72.07] | 48.03 [35.57 to 73.08] | 48.03 [47.77 to 72.07]

10. Secondary Outcome: Volume of Distribution at Steady State (Intravenous Dosing) (Vss/F) for the Analysis of PK Parameter
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Litre | 1275 (612.8) | 1190 (586.4) | 2756 (1577) | 1472 (855.9) | 1645 (1157)

11. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) for the Analysis of PK Parameter
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and up to 72-hour Post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Litre | 1529 (953.1) | 1490 (779.9) | 3120 (2066) | 1810 (1120) | 1719 (1608)

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: To assess AEs as variable of safety and tolerability of single doses of verinurad in healthy participants.
Time Frame: From screening (Day -28 to Day -2) till follow-up visit (7 to 14 days post-final dose)
Population: All subjects who received at least 1 dose of verinurad (any formulation) were included in the safety analysis for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Participants
  Any treatment emergent adverse event (TEAE) | 5 | 6 | 2 | 4 | 3
  Related TEAEs | 2 | 0 | 1 | 3 | 0
  Any serious TEAE (including death) | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to discontinuation of IMP | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to withdrawal from study | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening (Day -28 to Day -2) till follow-up visit (7 to 14 days post-final dose)
Arm/Group | Treatment 1: 1 x 12 mg ER8 Capsule Fasted | Treatment 2: 2 x 6 mg A-capsule Fasted | Treatment 3: 2 x 6 mg A-capsule Fed | Treatment 4: 2 x 6 mg B-capsule Fasted | Treatment 5: 2 x 6 mg B-capsule Fed
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 5/25 | 6/25 | 2/25 | 4/25 | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1: 1 x 12 mg ER8 Capsule Fasted (N=25) | Treatment 2: 2 x 6 mg A-capsule Fasted (N=25) | Treatment 3: 2 x 6 mg A-capsule Fed (N=25) | Treatment 4: 2 x 6 mg B-capsule Fasted (N=25) | Treatment 5: 2 x 6 mg B-capsule Fed (N=25)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This confidential document is the property of AstraZeneca AB. No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT04024501/Prot_SAP_000.pdf